CLINICAL TRIAL: NCT05714319
Title: Intracoronary Provocative Test With Acetylcholine in Patients With Stable Myocardial Ischemia or Myocardial Infarction and Non-Obstructive Coronary Arteries: the "Provoke" Study
Brief Title: Intracoronary Provocative Test With Acetylcholine in Patients With INOCA and MINOCA
Acronym: Provoke
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, MONTONE ROCCO ANTONIO, IRCCS Researcher, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5404
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Myocardial Infarction With Non-Obstructive Coronary Artery; Ischemia With Non-Obstructive Coronary Artery
Keywords: MINOCA; INOCA
MeSH Terms: conditions — MINOCA | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MINOCA: Patients undergoing clinically indicated CAG for suspected myocardial ischemia with angiographic evidence of non-obstructive CAD (angiographically normal coronary arteries or diffuse atherosclerosis with stenosis <50% and/or fractional flow reserve [FFR] >0.80 if coronary stenosis ranging from 40 to 49%) that underwent an intracoronary provocative test with ACh according to clinical practice and medical choice will be enrolled.
  Patients with MINOCA will be diagnosed based on clinical evidence of acute myocardial ischemia, detection of raise and fall of serum troponin T levels with at least one value exceeding the 99th percentile of a normal reference population and at least one of the following: myocardial ischemia (1 or + episodes of chest pain at rest typical enough to suggest a cardiac ischemic origin in the previous 24 hours); new ischemic ECG changes; pathological Q waves; new loss of viable myocardium or regional wall motion abnormality consistent with an ischemic aetiology.
  Interventions: Other: Data collection; Other: Clinical follow-up
- INOCA: All consecutive patients undergoing clinically indicated CAG for suspected myocardial ischemia with angiographic evidence of non-obstructive CAD (angiographically normal coronary arteries or diffuse atherosclerosis with stenosis <50% and/or fractional flow reserve [FFR] >0.80 if coronary stenosis ranging from 40 to 49%) that underwent an intracoronary provocative test with ACh as suggested in current guidelines and consensus and according to clinical practice and medical choice will be consecutively included in this study.
  Patients with INOCA will be defined as those with a stable pattern of typical chest pain on exertion, at rest or both, without any sign of acute myocardial infarction (MI), and/or evidence of inducible myocardial ischemia undergoing a scheduled hospital admission for CAG.
  Interventions: Other: Data collection; Other: Clinical follow-up

INTERVENTIONS:
Other: Data collection — Variables collected will include:
  * demographics (sex, age)
  * comorbidities (type 2 diabetes mellitus, familiar history of CAD, smoke habit, dyslipidaemia, hypertension, history of CAD)
  * echocardiographic (left ventricle ejection fraction at admission, the presence and grade of diastolic dysfunction, and the presence and grade of any valvulopathies)
  * angiographic data (presence of non-obstructive CAD (any coronary lesion <50% diameter stenosis), the presence of myocardial bridge and, if this latter is present, its localization and length)
  * laboratory measurements (hematologic variables (haemoglobin and white blood cells), creatinine, high sensitivity cardiac troponin I (hs-cTnI), and C-reactive protein (CRP) at the time of admission)
  * medical therapy at admission
  * response to intracoronary provocative test with ACh.
Other: Clinical follow-up — All patients will undergo a clinical follow-up by telephonic interview and/or clinical visit at 6, 12, 24, 36, 48 and 60 months from hospital discharge, during which the incidence of MACCE in the past months will be investigated and collected.

SUMMARY:
Coronary vasomotor disorders, occurring both at microvascular and epicardial level, have been demonstrated as responsible for myocardial ischemia in a sizeable group of patients undergoing coronary angiography (CAG), with clinical manifestations ranging from ischemia with non-obstructive coronary arteries (INOCA) to myocardial infarction with non-obstructive coronary arteries (MINOCA), along with life-threatening arrhythmias and sudden cardiac death. Intracoronary provocative testing with administration of acetylcholine (ACh) at the time of CAG may elicit epicardial coronary spasm or microvascular spasm in susceptible individuals, and therefore is assuming paramount importance for the diagnosis of functional coronary alterations in patients with suspected myocardial ischemia and non-obstructive coronary artery disease (CAD). However, previous studies mainly focused on patients with INOCA, whilst MINOCA patients were often underrepresented. Assessing the presence of coronary vasomotor disorders is of mainstay importance in order to implement the optimal management and improve clinical outcomes. Clinical predictors for a positive ACh test could allow the development of predictive models for a positive or negative response based on clinical and/or angiographic features readily available in the catheterization laboratories, thus helping clinicians in the diagnosis of coronary vasomotor disorders even in patients at high risk of complications.

DETAILED DESCRIPTION:
Background

Coronary vasomotor disorders, occurring both at microvascular and epicardial level, have been demonstrated as responsible for myocardial ischemia in a sizeable group of patients undergoing coronary angiography (CAG), with clinical manifestations ranging from ischemia with non-obstructive coronary arteries (INOCA) to myocardial infarction with non-obstructive coronary arteries (MINOCA), along with life-threatening arrhythmias and sudden cardiac death. Intracoronary provocative testing with administration of acetylcholine (ACh) at the time of CAG may elicit epicardial coronary spasm or microvascular spasm in susceptible individuals, and therefore is assuming paramount importance for the diagnosis of functional coronary alterations in patients with suspected myocardial ischemia and non-obstructive coronary artery disease (CAD). However, previous studies mainly focused on patients with INOCA, whilst MINOCA patients were often underrepresented . In addition, intracoronary provocative testing is still largely underused in clinical practice, probably because of concerns regarding the risk of complications, especially in the acute clinical setting. Of note, the landmark "Coronary Microvascular Angina" (CorMicA) trial demonstrated that a strategy of adjunctive invasive testing for disorders of coronary function in patients with non-obstructive CAD linked with stratified medical therapy is superior to usual care in improving patients' outcomes, including reduction in angina severity and better quality of life. Therefore, assessing the presence of coronary vasomotor disorders is of mainstay importance in order to implement the optimal management and improve clinical outcomes.

Of interest, the investigators recently demonstrated that performing an ACh provocative test in patients with myocardial ischemia and non-obstructive coronary arteries is safe with a low rate of complications, without differences between patients presenting with INOCA or MINOCA. In particular, a previous history of paroxysmal atrial fibrillation (AF), a moderate-to-severe left ventricle (LV) diastolic dysfunction and a higher corrected QT (QTc) dispersion at baseline electrocardiogram (ECG) were independent predictors for the occurrence of complications during the test and, therefore, patients with these characteristics may be those requiring particular attention during the test. Moreover, the investigators demonstrated that performing an ACh provocative test has relevant prognostic implications, as patients with a positive test have a higher risk of major adverse cerebrovascular and cardiovascular events (MACCE) at follow-up, and, therefore, performing an ACh test can help in stratifying the prognosis, especially in MINOCA patients, suggesting the presence of a net clinical benefit deriving from its use. Furthermore, the investigators recently demonstrated that some clinical (MINOCA as clinical presentation and elevated circulating levels of C-reactive protein) and angiographic (presence of myocardial bridging) features are independent predictors for a positive response to ACh test.

Of interest, the identification of clinical predictors for a positive ACh test could allow the development of predictive models for a positive or negative response based on clinical and/or angiographic features readily available in the catheterization laboratories, thus helping clinicians in the diagnosis of coronary vasomotor disorders even in patients at high risk of complications (e.g.: history of AF, LV diastolic dysfunction, long QTc interval or QTc dispersion at baseline ECG, bradyarrhythmia). Moreover, the implementation of such predictive models in clinical practice could avoid the need of performing a provocative test, significantly reducing the duration of invasive procedures as well as the associated risks and allowing a fast determination of the most appropriate treatments and clinical paths, an efficient planning, and a parsimonious use of medical resources. In addition, developing predictive models for the risk of future cardiovascular events could help clinicians in the prognostic stratification and the choice of therapeutic strategies in the post-discharge management, possibly identifying those patients that may need a more aggressive therapy and a closer follow-up.

Therefore, the investigators hypothesize that:

* Clinical predictors for a positive ACh test response could be identified, allowing the development of predictive models and/or clinical risk scores that could help clinicians in the diagnosis of coronary vasomotor disorders and the implementation of the most appropriate management.
* A positive ACh test could be associated with a higher rate of adverse cardiovascular events at follow-up, thus helping in the prognostic stratification of INOCA and MINOCA patients and identifying those that may need a more aggressive therapy and a closer follow-up.

Primary objective

To derive and validate predictive models/clinical risk scores able to predict a positive ACh test response in INOCA and MINOCA patients basing on clinical and/or angiographic features.

Secondary objective

To derive and validate predictive models/clinical risk scores able to predict a worse clinical outcome in terms of major adverse cardiovascular and cerebrovascular events (MACCE), defined as the composite of cardiovascular death, nonfatal myocardial infarction (MI), hospitalization due to unstable angina (UA), and stroke/transient ischemic attack (TIA) in INOCA and MINOCA patients basing on clinical and/or angiographic features.

Study design

Observational study.

Sample size calculation

Up to our knowledge no study has investigated the creation of a potential score for Ach test positivity. Hence this would represent the first and, as such, is includable among pilot studies and, therefore, no formal sample size calculation is needed, but all of patients satisfying inclusion criteria can be included. Based on the study design, which pertains the creation and validation of a score, which would require a training and validation cohort, and will alongside imply the use of regression methods, the investigators plan to include 600 patients. Such a sample size would allow for the stratification in two cohort and the analysis of the approximately 50 covariates included in the study. In fact, according to van Smeden, events per variable (EPV) may go beyond the common rule of EPV≥10.

Statistical analysis

Descriptive analysis and between-groups comparisons

The sample will be described in its demographic, anthropometric, clinical, instrumental, variables through descriptive statistical techniques. In depth, qualitative variables will be expressed by absolute and relative percentage frequencies. Quantitative variables, indeed, will be reported either as mean and standard deviation (SD) or median and interquartile range (IQR), respectively in the case they were normally or not normally distributed. Their distribution will be previously assessed by the Shapiro Wilk test. Between groups differences in the demographic, clinical, laboratory and pathologic features will be assessed by the Chi Square or the Fisher's exact test as for qualitative variables (with Freeman- Halton's extension when appropriate), whilst quantitative variables will be evaluated either by the Student's t test or the Mann- Withney U test, according to their distribution.

Derivation and validation of clinical risk scores

Data used for score development will be derived from a prospectively enrolled sample of 550 NOCAD patients, consecutively admitted to the Department of Cardiovascular Sciences of Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome (Italy). There is no generally accepted approach for the estimation of the sample size for derivation of score prediction models. Hence, the investigators based for the derivation of the score to include in the multivariable model a number of covariates consistent with the most recent rules on the minimum number of events per variable needed. The investigators will randomly allocate the participants to two cohorts, one cohort will be used to develop the score model (derivation cohort), and the other to validate and assess the diagnostic abilities of the score (validation cohort). Multiple imputation will be applied to handle missing data, by "imputeR" R package. Univariable and multivariable regression models will be performed on the derivation cohort to identify independent predictors of a positive ACh test to be included in the scoring system. In depth, the investigators will compute Odd Ratios (ORs) and 95% Confidence Intervals (CIs) of the predictor candidates for the outcome (i.e., positive Ach test) by univariable logistic regression models. Predictors to be included in the multivariable model will be selected based on univariable analysis (p<0.05 or suggestive, i.e. 0.05<p<0.10) and expert opinion. The multivariable logistic regression model will produce β coefficient and Standard Errors (SE) for each variable. The performance of the model will be assessed based on diverse methods, such as Somers' Dxy rank correlation, C-index, Nagelkerke R2 value, calibration intercept and slope, and Brier score. Finally, the Hosmer-Lemeshow goodness-of-fit test will allow for the calibration in the derivation cohort. Calibration plots will further provide a graphic representation of the association between the predicted and observed outcome by locally weighted scatterplot smoothing. "rms", "predtools" and "magrittr" R packages will be used for the whole analyses set. Internal validation of the model will be performed based on a bootstrap procedure. The investigators will then pass to develop a scoring system to predict the outcome providing an integer value to each predictor included in the scoring system based on each variable's β coefficient in the derivation cohort. Appropriate cutoff values will be set for a rule-in and rule-out approach to help in decision-making. In depth, quantitative independent predictors will be further transformed into either ordinal or nominal qualitative variables. Transformation will be performed seeking for one or more optimal cut-points by appropriate selection methods based on ROC curves analysis, by mean of "pROC" R package. Particularly, "OptimalCutpoints" R package will be used applying the SpEqualSe selection method, which returns the highest accuracy. The diagnostic abilities (i.e., sensitivity, specificity, positive likelihood ratio, and negative likelihood ratio) of each score will be then calculated, and the patients will be divided into 3 groups (positive, negative, suspect). For validation, the developed score will be applied to the validation cohort, and the discrimination and calibration performances will be described, as aforementioned. The overall performance will be described in terms of Sensitivity, Specificity, Accuracy (or Positive Predictive Value, PPV), F1 Score, Accuracy, False Positive Rate (FPR), False Discovery Rate (FDR) and False Negative Rate (FNR). Statistical analyses will be carried out using R software, version 4.2.0 (CRAN ®, R Core 2022).

Derivation and validation of predictive models using artificial intelligence/machine learning models (second phase)

In the second phase of this study, the investigators further plan to develop a predictive model of MACCE in the studied population, as well as to extend the study out of our clinical facility to potentially validate the models also externally. In this context, the investigators foresee to further enhance the analysis by adding Machine Learning methods, such as XGBoost, Random Forest, Neural Networks, which will be chosen based on the type of data and question to be answered. ML methods will be applied in Python software.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* INOCA or MINOCA as clinical presentation.
* Patient that underwent an intracoronary provocative test with ACh at the time of CAG, as suggested in current guidelines and consensus and according to clinical practice and medical choice and independently from the present study.
* Patients with INOCA will be defined as those with a stable pattern of typical chest pain on exertion, at rest or both, without any sign of acute myocardial infarction (MI), and/or evidence of inducible myocardial ischemia undergoing a scheduled hospital admission for CAG.
* Patients with MINOCA will be diagnosed based on clinical evidence of acute myocardial ischemia, detection of raise and fall of serum troponin T levels with at least one value exceeding the 99th percentile of a normal reference population and at least one of the following: 1) symptoms of myocardial ischemia (one or more episodes of chest pain at rest typical enough to suggest a cardiac ischemic origin in the previous 24 hours); 2) new ischemic ECG changes (ST-segment and/or T wave abnormalities); 3) development of pathological Q waves; 4) imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic aetiology (19).
* Written informed consent to participate.

Exclusion Criteria:

* Patient that did not undergo an intracoronary provocative test with ACh at the time of CAG.
* Among patients presenting with suspected MINOCA, those with obvious causes of MI other than suspected coronary vasomotor abnormalities will be excluded (e.g.: Takotsubo syndrome, suspected diagnosis of myocarditis, pulmonary embolism, evidence of coronary thrombosis on an unstable plaque confirmed by optical coherence tomography, cardiotoxic drug administration, hypertensive crisis or severe valvulopathies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Department of Cardiovascular Sciences of Fondazione Policlinico Universitario A. Gemelli IRCCS since January 1, 2020 undergoing clinically indicated CAG for suspected myocardial ischemia with angiographic evidence of non-obstructive CAD (angiographically normal coronary arteries or diffuse atherosclerosis with stenosis <50% and/or fractional flow reserve [FFR] >0.80 if coronary stenosis ranging from 40 to 49%) that underwent an intracoronary provocative test with ACh as suggested in current guidelines and consensus and according to clinical practice and medical choice will be consecutively included in this study. Both patients admitted with suspected INOCA and MINOCA, diagnosed according to the most recent guidelines, will be enrolled.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2027-06-12 (Estimated); Study Completion 2028-01-12 (Estimated)

PRIMARY OUTCOMES:
Assess clinical predictors for a positive ACh test response | Up to 30 days
  To assess for the presence of clinical predictors for a positive ACh test response in INOCA and MINOCA patients that could be used to develop and validate predictive models and/or clinical risk scores for a positive ACh test.

SECONDARY OUTCOMES:
Assess clinical predictors for MACCE | Up to 2 years
  To assess for the presence of clinical predictors for MACCE in INOCA and MINOCA patients that could be used to develop and validate predictive models and/or clinical risk scores for MACCE at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco A Montone, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maseri A, Severi S, Nes MD, L'Abbate A, Chierchia S, Marzilli M, Ballestra AM, Parodi O, Biagini A, Distante A. "Variant" angina: one aspect of a continuous spectrum of vasospastic myocardial ischemia. Pathogenetic mechanisms, estimated incidence and clinical and coronary arteriographic findings in 138 patients. Am J Cardiol. 1978 Dec;42(6):1019-35. doi: 10.1016/0002-9149(78)90691-4. No abstract available. PMID 727129
- [Background] Inami T, Kataoka M, Shimura N, Ishiguro H, Kohshoh H, Taguchi H, Yanagisawa R, Hara Y, Satoh T, Yoshino H. Left ventricular dysfunction due to diffuse multiple vessel coronary artery spasm can be concealed in dilated cardiomyopathy. Eur J Heart Fail. 2012 Oct;14(10):1130-8. doi: 10.1093/eurjhf/hfs103. Epub 2012 Jun 19. PMID 22713288
- [Background] Ong P, Aziz A, Hansen HS, Prescott E, Athanasiadis A, Sechtem U. Structural and Functional Coronary Artery Abnormalities in Patients With Vasospastic Angina Pectoris. Circ J. 2015;79(7):1431-8. doi: 10.1253/circj.CJ-15-0520. Epub 2015 Jun 18. PMID 26084380
- [Background] Montone RA, Niccoli G, Fracassi F, Russo M, Gurgoglione F, Camma G, Lanza GA, Crea F. Patients with acute myocardial infarction and non-obstructive coronary arteries: safety and prognostic relevance of invasive coronary provocative tests. Eur Heart J. 2018 Jan 7;39(2):91-98. doi: 10.1093/eurheartj/ehx667. PMID 29228159
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Montone RA, Meucci MC, De Vita A, Lanza GA, Niccoli G. Coronary provocative tests in the catheterization laboratory: Pathophysiological bases, methodological considerations and clinical implications. Atherosclerosis. 2021 Feb;318:14-21. doi: 10.1016/j.atherosclerosis.2020.12.008. Epub 2020 Dec 13. PMID 33360263
- [Background] Niccoli G, Morrone D, De Rosa S, Montone RA, Polimeni A, Aimo A, Mancone M, Muscoli S, Pedrinelli R, Indolfi C; Interventional Cardiology and the Coronary Pathophysiology and Microcirculation Study Groups of the Italian Society of Cardiology, and on behalf of the Italian Society of Cardiology. The central role of invasive functional coronary assessment for patients with ischemic heart disease. Int J Cardiol. 2021 May 15;331:17-25. doi: 10.1016/j.ijcard.2021.01.055. Epub 2021 Jan 30. No abstract available. PMID 33529656
- [Background] Ong P, Athanasiadis A, Borgulya G, Vokshi I, Bastiaenen R, Kubik S, Hill S, Schaufele T, Mahrholdt H, Kaski JC, Sechtem U. Clinical usefulness, angiographic characteristics, and safety evaluation of intracoronary acetylcholine provocation testing among 921 consecutive white patients with unobstructed coronary arteries. Circulation. 2014 Apr 29;129(17):1723-30. doi: 10.1161/CIRCULATIONAHA.113.004096. Epub 2014 Feb 26. PMID 24573349
- [Background] Probst S, Seitz A, Martinez Pereyra V, Hubert A, Becker A, Storm K, Bekeredjian R, Sechtem U, Ong P. Safety assessment and results of coronary spasm provocation testing in patients with myocardial infarction with unobstructed coronary arteries compared to patients with stable angina and unobstructed coronary arteries. Eur Heart J Acute Cardiovasc Care. 2020 Jun 8:2048872620932422. doi: 10.1177/2048872620932422. Online ahead of print. PMID 33609124
- [Background] Zaya M, Mehta PK, Merz CN. Provocative testing for coronary reactivity and spasm. J Am Coll Cardiol. 2014 Jan 21;63(2):103-9. doi: 10.1016/j.jacc.2013.10.038. Epub 2013 Nov 6. PMID 24201078
- [Background] Agewall S, Beltrame JF, Reynolds HR, Niessner A, Rosano G, Caforio AL, De Caterina R, Zimarino M, Roffi M, Kjeldsen K, Atar D, Kaski JC, Sechtem U, Tornvall P; WG on Cardiovascular Pharmacotherapy. ESC working group position paper on myocardial infarction with non-obstructive coronary arteries. Eur Heart J. 2017 Jan 14;38(3):143-153. doi: 10.1093/eurheartj/ehw149. No abstract available. PMID 28158518
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- [Background] Montone RA, Rinaldi R, Del Buono MG, Gurgoglione F, La Vecchia G, Russo M, Caffe A, Burzotta F, Leone AM, Romagnoli E, Sanna T, Pelargonio G, Trani C, Lanza GA, Niccoli G, Crea F. Safety and prognostic relevance of acetylcholine testing in patients with stable myocardial ischaemia or myocardial infarction and non-obstructive coronary arteries. EuroIntervention. 2022 Oct 7;18(8):e666-e676. doi: 10.4244/EIJ-D-21-00971. PMID 35377315
- [Background] Montone RA, Gurgoglione FL, Del Buono MG, Rinaldi R, Meucci MC, Iannaccone G, La Vecchia G, Camilli M, D'Amario D, Leone AM, Vergallo R, Aurigemma C, Buffon A, Romagnoli E, Burzotta F, Trani C, Crea F, Niccoli G. Interplay Between Myocardial Bridging and Coronary Spasm in Patients With Myocardial Ischemia and Non-Obstructive Coronary Arteries: Pathogenic and Prognostic Implications. J Am Heart Assoc. 2021 Jul 20;10(14):e020535. doi: 10.1161/JAHA.120.020535. Epub 2021 Jul 14. PMID 34259010
- [Background] Kunadian V, Chieffo A, Camici PG, Berry C, Escaned J, Maas AHEM, Prescott E, Karam N, Appelman Y, Fraccaro C, Louise Buchanan G, Manzo-Silberman S, Al-Lamee R, Regar E, Lansky A, Abbott JD, Badimon L, Duncker DJ, Mehran R, Capodanno D, Baumbach A. An EAPCI Expert Consensus Document on Ischaemia with Non-Obstructive Coronary Arteries in Collaboration with European Society of Cardiology Working Group on Coronary Pathophysiology & Microcirculation Endorsed by Coronary Vasomotor Disorders International Study Group. Eur Heart J. 2020 Oct 1;41(37):3504-3520. doi: 10.1093/eurheartj/ehaa503. PMID 32626906
- [Background] Ford TJ, Ong P, Sechtem U, Beltrame J, Camici PG, Crea F, Kaski JC, Bairey Merz CN, Pepine CJ, Shimokawa H, Berry C; COVADIS Study Group. Assessment of Vascular Dysfunction in Patients Without Obstructive Coronary Artery Disease: Why, How, and When. JACC Cardiovasc Interv. 2020 Aug 24;13(16):1847-1864. doi: 10.1016/j.jcin.2020.05.052. PMID 32819476
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Background] Beltrame JF, Crea F, Kaski JC, Ogawa H, Ong P, Sechtem U, Shimokawa H, Bairey Merz CN; Coronary Vasomotion Disorders International Study Group (COVADIS). International standardization of diagnostic criteria for vasospastic angina. Eur Heart J. 2017 Sep 1;38(33):2565-2568. doi: 10.1093/eurheartj/ehv351. PMID 26245334
- [Background] Ong P, Camici PG, Beltrame JF, Crea F, Shimokawa H, Sechtem U, Kaski JC, Bairey Merz CN; Coronary Vasomotion Disorders International Study Group (COVADIS). International standardization of diagnostic criteria for microvascular angina. Int J Cardiol. 2018 Jan 1;250:16-20. doi: 10.1016/j.ijcard.2017.08.068. Epub 2017 Sep 8. PMID 29031990
- [Background] van Smeden M, Moons KG, de Groot JA, Collins GS, Altman DG, Eijkemans MJ, Reitsma JB. Sample size for binary logistic prediction models: Beyond events per variable criteria. Stat Methods Med Res. 2019 Aug;28(8):2455-2474. doi: 10.1177/0962280218784726. Epub 2018 Jul 3. PMID 29966490
- [Background] Moons KG, Altman DG, Reitsma JB, Ioannidis JP, Macaskill P, Steyerberg EW, Vickers AJ, Ransohoff DF, Collins GS. Transparent Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis (TRIPOD): explanation and elaboration. Ann Intern Med. 2015 Jan 6;162(1):W1-73. doi: 10.7326/M14-0698. PMID 25560730